CLINICAL TRIAL: NCT04383964
Title: Transport Distraction Osteogenesis for Reconstruction of Ramus-Condyle Unit Following Release of Temporomandibular Joint Ankylosis
Brief Title: Transport Distraction Osteogenesis for Ramus-Condyle Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Distraction Osteogenesis
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Bilateral or Unilateral Deficient Ramus-condyle Unit
MeSH Terms: interventions — Osteogenesis, Distraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transport distraction osteogenesis (Experimental): Locally made and designed submerged monodirectional in the vertical (Y) axis distractor was used.
  A transport disc is created at the remaining stump of the RCU with an L shaped osteotomy.
  The prepared disc is to be wide enough to fit the upper portion of the distrcator.
  The submerged distractor will be placed in a position to guide the transport disc moving up and backwards toward the glenoid fossa.
  The length of the distractor is determined according to the amount of distraction planned to reach the glenoid fossa.
  Interventions: Device: Distraction Osteogenesis for Reconstruction of Ramus-Condyle

INTERVENTIONS:
Device: Distraction Osteogenesis for Reconstruction of Ramus-Condyle — transport distraction osteogenesis in restoring the deficient condyle/ramus unit of patients with TMJ ankylosis to correct the resultant deformity either unilaterally or bilaterally.

SUMMARY:
this study was done to evaluate the use of transport distraction osteogenesis in restoring the deficient condyle/ramus unit of patients with unilateral or bilateral TMJ ankylosis to correct the resultant deformity

DETAILED DESCRIPTION:
10 patients with post ankylosis deficient ramus /condyle unit who underwent release procedure in the Maxillofacial and Plastic Surgery Department, Faculty of Dentistry, Alexandria University, Egypt.

all patients were assessed clinically and by imaging using OPG, lateral and PA cephalometry, and cone beam CT to assess the deficient ramus/condyle unit (RCU) then patients were operated using transport distraction osteogenesis to lengthen the RCU. Then follow up of all patients both clinically and radiographically was adopted.

ELIGIBILITY:
Inclusion Criteria:

* Post ankylosis deformity: Bilateral or unilateral deficient ramus-condyle unit (RCU) after TMJ release

Exclusion Criteria:

* Mentally affected patients.
* Medically compromised patients.
* Post menopausal osteoporosis.

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Jaw movements (changes in jaw movements through 18 months follow up) | at 3rd, 6th and 18th months
  Mouth opening in mm, Jaw movement in lateral excursion and opening.
Ramus height (changes of ramus heights through 18 months follow up) | at 3rd and 6th months
  Determination of the height of the ramus by PA cephalometric, Lateral cephalometric x-rays and tracings

SECONDARY OUTCOMES:
Occlusal discrepancy or anterior open bite | 18th months
  Occlusal discrepancy or anterior open bite

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria, Azarita, Egypt